CLINICAL TRIAL: NCT06320457
Title: Supporting People Involuntarily Admitted to a Psychiatric Hospital Through a Brief Case Management Intervention That Promotes Personal Recovery and Reduces the Negative Effects of Coercion: a Pilot Study
Brief Title: A Brief Case Management Intervention for People Involuntarily Admitted to a Psychiatric Hospital
Acronym: CARP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Stéphane Morandi, Deputy Head of the Community Psychiatry Service, PD & MER, University of Lausanne Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-00095
Record Dates: First submitted 2024-03-04; First posted 2024-03-20 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Psychiatric Disorder; Involuntary Psychiatric Hospitalization
Keywords: coercion; involuntary admission; personal recovery; case management; psychiatry
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): Brief case management intervention group
  Interventions: Other: Brief case management intervention

INTERVENTIONS:
Other: Brief case management intervention — The brief case management intervention aims to support patients during the difficult phase of involuntary hospitalisation and reduce the impact of this short-term event on their long-term recovery process. The intervention starts during the hospital stay, at the latest one week after admission, and lasts for a maximum of one month after discharge. The intervention consists of five sessions, the order of which may vary according to the specific needs of the patient:
  1. Personal account of involuntary hospitalisation and its consequences
  2. Presentation of the personal recovery model and the tools to promote it and prevent coercion
  3. Introduction to the personal recovery plan
  4. Network meeting and discussion on "dignity of risk"
  5. Personal recovery plan

SUMMARY:
The goal of this clinical trial is to assess whether a brief case management intervention aimed at promoting personal recovery and reducing the negative effects of coercion among people involuntarily admitted to a psychiatric hospital would be well accepted by them, practically feasible and useful. The main questions it aims to answer are:

* Is the case management intervention acceptable and feasible?
* What are the preliminary effects of the case management intervention on patients' personal recovery and its sub-dimensions, as well as on their level of perceived coercion and their global satisfaction with hospital care?

Participants will be asked to take part in:

* the five sessions of the case management intervention;
* two evaluation sessions (pre and post-intervention);
* a final in-depth semi-structured interview (optional).

ELIGIBILITY:
Inclusion Criteria:

* To have been involuntarily admitted by a medical doctor
* To be aged between 18 and 65 years

Exclusion Criteria:

* Patients unable to provide written consent due to a lack of discernment
* Patients unable to speak French well enough to participate in the study without the help of an interpreter

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Eligibility rate | From start of study recruitment through study recruitment completion, on average 6 months
  Number of eligible patients/number of patients involuntarily hospitalised on site during study period as reported in a structured flowchart by the case managers after each site visit
Participation rate | From start of study recruitment through study recruitment completion, on average 6 months
  Number of patients accepting to participate/number of approached patients as reported in a structured flowchart by the case managers after each site visit and based on the number of signed consent forms
Drop-out rate | Post-intervention, up to 1 month post hospital discharge
  Number of patients who completed the programme/number of recruited patients as reported by case managers in a structured questionnaire detailing which intervention sessions were delivered to each patient
Intervention dosage | Post-intervention, up to 1 month post hospital discharge
  Mean number of sessions delivered per participant as reported by case managers in a structured questionnaire detailing which intervention sessions were delivered to each patient
Missing data rates | At the end of the study, on average 9 months after the inclusion of the first participant
  Percentage of missing data
Number of unexpected adverse events | Up to 1 week after hospital admission through up to 1 month post hospital discharge
  Number of unexpected adverse events related to the intervention reported in a structured form by the case managers or the investigator
Participants' acceptance and degree of satisfaction | Post-intervention, up to 1 month post hospital discharge
  Participants' acceptance and degree of satisfaction with both the intervention and the research process qualitatively assessed through semi-structured interviews
Implementation barriers and facilitating factors | After the last included participant final evaluation, on average 8 months after the inclusion of the first participant
  Barriers and facilitating factors encountered throughout the implementation process as described by some members of the hospital team, during in-depth semi-structured interviews.

SECONDARY OUTCOMES:
Recovery Assessment Scale (RAS) | Two time points assessment: up to 1 week after hospital admission (pre-intervention) and up to 1 month post hospital discharge (post-intervention)
  The French validated version of the Recovery Assessment Scale (RAS), a 24-item, patient-oriented outcome inventory which assesses personal recovery on a five-point Likert scale ranging from 1="strongly disagree" to 5="strongly agree". The instrument provides a total score of personal recovery as well as sub-scores on five specific dimensions: personal confidence and hope, willingness to ask for help, goal and success orientation, reliance on others, no domination by symptoms. Both the total score and the five sub-scores are used in the study. Higher scores correspond to better recovery.
Empowerment Scale | Two time points assessment: up to 1 week after hospital admission (pre-intervention) and up to 1 month post hospital discharge (post-intervention)
  The validated Empowerment Scale, a 28-item measure assessing personal empowerment as defined by mental health service-users on a four-point Likert scale ranging from "strongly disagree" to "strongly agree". The total score is used for the study. Higher scores correspond to higher empowerment.
Rosenberg Self-Esteem Scale (RSS) | Two time points assessment: up to 1 week after hospital admission (pre-intervention) and up to 1 month post hospital discharge (post-intervention)
  The French validated version of the Rosenberg Self-Esteem Scale (RSS), a very short 10-item inventory measuring self-esteem on a four-point Likert scale from 1="strongly disagree" to 4="strongly agree". The RSS total score may range between 10 and 40, with higher scores indicating higher level of self-esteem.
The Paradox of Self-Stigma scale (PaSS-24) | Two time points assessment: up to 1 week after hospital admission (pre-intervention) and up to 1 month post hospital discharge (post-intervention)
  The Paradox of Self-Stigma scale (PaSS-24), a short French-language scale measuring self-stigma and its three related construct of stereotype endorsement, righteous anger and non-disclosure. It includes 24 items rated on a five-point Likert scale ranging between 1="strongly disagree" and 5="strongly agree". The three sub-scores are used in the study.
Beck Hopelessness Scale (BHS) | Two time points assessment: up to 1 week after hospital admission (pre-intervention) and up to 1 month post hospital discharge (post-intervention)
  The French validated version of the Beck Hopelessness Scale (BHS), an inventory of 20 true-false items which assess negative expectations about the future on three dimensions: feeling about the future, decrease in motivation and expectations. BHS total score can range between 0 and 20, with higher scores reflecting higher levels of hopelessness.
WHOQOL-BREF | Two time points assessment: up to 1 week after hospital admission (pre-intervention) and up to 1 month post hospital discharge (post-intervention)
  The French validated version of the WHOQOL-BREF, a scale including 26 Likert type items, measuring quality of life in four domains: physical health, psychological health, social relationships and environment. Its total score is used in the study.
International Trauma Questionnaire (ITQ) | Two time points assessment: up to 1 week after hospital admission (pre-intervention) and up to 1 month post hospital discharge (post-intervention)
  The French validated version of the International Trauma Questionnaire (ITQ), a scale to assess Post Traumatic Stress Disorder (PTSD) and Complex Post Traumatic Stress Disorder (C-PTSD) symptoms among adults. The inventory includes 18 items: six to assess the PTSD, six to assess the Disorders in Self Organisation (DSO), and six to assess functional impairment in several important areas of life. Respondents are required to indicate, on a five-point scale from 0="not at all" to 4="extremely", how much each symptom has bothered them in the past month. A total score, ranging between 0 and 24, can be calculated for the PTSD and DSO subscale. A C-PTSD score, ranging between 0 and 48, can also be calculated by adding the PTSD and DSO subscales. Both the PTSD and the C-PTSD total scores will be used in the study.
Coercion Ladder (CL) | Two time points assessment: up to 1 week after hospital admission (pre-intervention) and up to 1 month post hospital discharge (post-intervention)
  The Coercion Ladder (CL), a single-item instrument asking patients to rate their experience of care on a visual analogue scale ranging from 1="minimum use of coercion" to 10="maximum use of coercion".
Index of fairness and Index of effectiveness | Two time points assessment: up to 1 week after hospital admission (pre-intervention) and up to 1 month post hospital discharge (post-intervention)
  The Index of fairness and the Index of effectiveness, two self-administered inventories which assess if participants perceived the experienced treatment pressures as fair and effective. The indices include four items each, rated on a five-point Likert scale from 1="strongly disagree" to 5="strongly agree". The two indices total scores are used in the study. Higher scores indicate higher perceived fairness and effectiveness.
Satisfaction with hospital care | Two time points assessment: up to 1 week after hospital admission (pre-intervention) and up to 1 month post hospital discharge (post-intervention)
  The Satisfaction with hospital care questionnaire, a six-item tool developed by the Swiss National Association for Quality Development in hospitals and clinics (ANQ), assessing patients' satisfaction about quality of treatment, information and communication, medication, patient's implication and discharge preparation, on a five-point Likert scale. The total score of global satisfaction is used in the study. Higher score corresponds to higher satisfaction. Moreover, the ANQ questionnaire includes one-item subscale on five-point assessing répondeurs' self-reported health. This subscale is also used in the study.
Brief INSPIRE scale | Post-intervention, up to 1 month post hospital discharge
  The Brief INSPIRE scale, a service user-rated measure assessing perceived staff support for personal recovery. The Brief INSPIRE consists of five items, one for each personal recovery domain. Responders are asked to rate on a five-point Likert scale, from 0="not at all" to 4="very much", how much they feel supported by staff in each domain of their personal recovery. A total score between 0 and 100 can be computed, with higher scores indicating higher perceived support.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Bonsack, Study Chair — Centre Hospitalier Universitaire Vaudois, CHUV
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No